CLINICAL TRIAL: NCT06436677
Title: A Study of Molecular Subtyping-based Therapeutic Strategies for Cutaneous T-cell Lymphoma
Acronym: AMITY
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Third Hospital (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Yang WANG, The Chief of Department of Dermatology and Venereology, Peking University First Hospital
Other Study IDs: PKU2024162-002; SF2024-1-4074 (Other Grant/Funding Number: Capital's Funds for Health Improvement and Research)
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Cutaneous T-Cell Lymphoma/Mycosis Fungoides; Cutaneous T Cell Lymphoma
Keywords: cutaneous T-cell lymphoma; mycosis fungoides; Sezary syndrome
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous; Sezary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Formalin fixed and paraffin embedded skin biopsy tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective study group: The group included patients with confirmed cutaneous T-cell lymphoma (CTCL) based on clinical features and histopathology from three research units: Peking University First Hospital, Peking University Third Hospital, and Beijing Institute of Cancer Prevention and Treatment. According to the immunohistochemistry algorithm established previously, the formalin-fixed and paraffin-embedded skin lesions of the patients will be stained. Patients will be assigned to different molecular subtypes, and the treatment strategy will be selected based on the classification.
  Interventions: Other: molecular subtype based treatment
- Retrospective control group: The control group included patients with complete baseline information and previous follow-up data in the TACTICAL database, established by Peking University First Hospital in 2009 for cutaneous lymphoma cases.

INTERVENTIONS:
Other: molecular subtype based treatment — The immunohistochemistry algorithm established by the previous research group was used to determine the molecular subtype, and the corresponding treatment plan was selected according to the subtype. Such as for TCyEM patients, interferon-based immunomodulatory therapy was selected, and TCM-type patients were treated with retinoids.
  Groups: Prospective study group

SUMMARY:
Cutaneous T-cell lymphoma (CTCL) is a group of diseases resulting from clonal hyperplasia of memory T cells in the skin. The increasing incidence and high treatment costs have posed significant challenges to public health and the economy. Current treatment guidelines only provide partial control, leading to varying remission times and recurrence rates. This study aims to use molecular subtyping and immunohistochemistry to guide treatment selection for CTCL patients, aiming to prolong clinical benefit, improve treatment safety, and reduce economic burden.

DETAILED DESCRIPTION:
The study focuses on the impact of treatment strategy selection based on molecular typing for patients with cutaneous T-cell lymphoma. The study aims to evaluate the effect on clinical benefit time and long-term prognosis, assess the safety of the treatment strategy, and explore the interaction between baseline factors and treatment regimens. This research could potentially provide valuable evidence for precision treatment in the context of cutaneous T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Patients with CTCL who do not respond well to targeted skin therapy (topical corticosteroids, nitrogen mustard, or phototherapy) in the early stage (stage I-IIA) and advanced stage (stage IIB-IV);
* Age 18-75 years;
* Expected survival time greater than 3 months (follow-up for the historical control group was greater than 3 months);

Exclusion Criteria:

* Received other anti-tumor therapy other than skin-targeted therapy (phototherapy, topical hormones or nitrogen mustard) within the past 1 month prior to enrollment;
* Patients with 2 or more types of primary cutaneous T-cell lymphoma at the same time;
* Combined with other malignant tumors, still receiving anti-tumor therapy;
* Has any other active disease that may increase the risk of protocol therapy or impair the patient's ability to receive protocol therapy, including but not limited to:

  * Comorbid epilepsy;
  * Comorbid autoimmune diseases;
  * Combined with hepatic decompensation;
  * Patients with renal insufficiency and creatinine clearance < 50ml/min;
* Have an uncontrollable medical condition, including but not limited to:

  * Ongoing or active infection;
  * Clinically significant healing or non-healing wounds;
  * Symptomatic congestive heart failure, unstable angina, clinically significant arrhythmias;
  * Significant lung disease (e.g., shortness of breath at rest or light activity, or need for supplemental oxygen for any reason);
  * Diseases/conditions that affect study compliance, such as infectious diseases or psychiatric illnesses/social situations, that are uncontrollable;
* Pregnant (or intending to become pregnant within 2 years) or lactating females;
* Concomitant participation in interventional clinical trials of other clinical trial drugs, except for questionnaire surveys or observational studies;
* Any situation in which the programme is not in compliance;
* Other conditions that in the opinion of the investigator are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, retrospective controls were selected from patients with complete baseline information and previous follow-up information in the cutaneous lymphoma case registry system (TACTICAL database) established in 2009. The prospective study group was a prospective enrollment of patients who met the inclusion criteria, and the immunohistochemistry algorithm established by the previous research group was used to determine the molecular subtype. The corresponding treatment regimen was selected according to the subtype. Follow-up was conducted according to the study design and updated by the ISCL, USCLC, and EORTC (2022) as they evaluate treatment response in patients. The primary outcome was time to clinical benefit (TTNT) of first-line therapy, defined as the time from treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
time to next treatment (TTNT) | From enrollment to the end of treatment at 2 years
  The time to treatment failure (TTNT) is defined as the duration from the start of treatment to when the treatment is switched to the next systemic therapy or until the patient passes away. Introducing new skin-directed therapy (SDT) alongside topical therapy doesn't indicate treatment failure unless the systemic treatment is changed. If the skin lesion worsens and needs local radiotherapy, it's considered that the systemic therapy has failed. The date of discontinuation of systemic therapy is used when treatment is stopped due to disease progression without further treatment.

SECONDARY OUTCOMES:
objective response rate (ORR) | From enrollment to the end of treatment at 2 years
  The objective response rate (ORR) is defined as the proportion of patients with complete response (CR) and partial response (PR) as per the Primary cutaneous lymphoma: recommendations for clinical trial design and staging update from the ISCL, USCLC, and EORTC (2022). The first CR or PR is achieved and repeated after 4 weeks for confirmation.
time to response (TTR) | From enrollment to the end of treatment at 2 years
  Time to response (TTR) is defined as the duration from the start of treatment to the first meeting of CR or PR criteria.
progression-free survival (PFS) | From enrollment to the end of treatment at 2 years
  The progression-free survival (PFS) is defined as the period from the beginning of treatment until the first instance of disease progression or death from any cause. Disease progression is defined as advancement to a higher TNMB stage (excluding changes from T1a or T2a to T1b or T2b) or death due to the disease.
overall survival (OS) | From enrollment to the end of treatment at 2 years
  The overall survival (OS) is defined as the period from the beginning of treatment to the point of death from any cause.

OTHER OUTCOMES:
adverse events and adverse effects | From enrollment to the end of treatment at 2 years
  Adverse events and adverse effects: The Preferred Term (PT) for adverse events and the Systemic Organ Classification (SOC) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). For the statistics of adverse event rates, each patient will be counted at most once per SOC and per PT. For the same adverse event that occurs multiple times in the same patient, the severity will be counted according to the severity of multiple occurrences. All adverse events (pre- and intra-treatment adverse events) are included in the list of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: YANG WANG, MD, Principal Investigator — Peking University First Hospital
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared within the participating medical units in the study, including study protocol, informed consent form, clinical study report and statistical analysis plan. Any other institutes requesting for IPD needs to be reviewed by the National Clinical Center for Skin and Immune Diseases in China.

REFERENCES:
- [Result] Olsen EA, Whittaker S, Willemze R, Pinter-Brown L, Foss F, Geskin L, Schwartz L, Horwitz S, Guitart J, Zic J, Kim YH, Wood GS, Duvic M, Ai W, Girardi M, Gru A, Guenova E, Hodak E, Hoppe R, Kempf W, Kim E, Lechowicz MJ, Ortiz-Romero P, Papadavid E, Quaglino P, Pittelkow M, Prince HM, Sanches JA, Sugaya M, Vermeer M, Zain J, Knobler R, Stadler R, Bagot M, Scarisbrick J. Primary cutaneous lymphoma: recommendations for clinical trial design and staging update from the ISCL, USCLC, and EORTC. Blood. 2022 Aug 4;140(5):419-437. doi: 10.1182/blood.2021012057. PMID 34758074
- [Result] Chen Z, Lin Y, Qin Y, Qu H, Zhang Q, Li Y, Wen Y, Sun J, Tu P, Gao P, Wang Y. Prognostic Factors and Survival Outcomes Among Patients With Mycosis Fungoides in China: A 12-Year Review. JAMA Dermatol. 2023 Oct 1;159(10):1059-1067. doi: 10.1001/jamadermatol.2023.2634. PMID 37585188